CLINICAL TRIAL: NCT05106335
Title: A Randomized, Open-Label, Controlled, Multi-Center Phase III Clinical Study of Camrelizumab Combined With Famitinib Malate Versus Docetaxel in Patients With Advanced Non-Small Cell Lung Cancer Who Progressed on Prior Immune Checkpoint Inhibitor Treatment and Platinum-Based Chemotherapy
Brief Title: A Study to Evaluate Camrelizumab Combined With Famitinib as Subsequent Therapy in Patients With Advanced NSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-332
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Advanced NSCLC
MeSH Terms: interventions — camrelizumab; famitinib; Docetaxel

STUDY DESIGN:
Intervention Model Description: Camrelizumab Combined with Famitinib Malate Versus Docetaxel
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm A (Experimental): camrelizumab + famitinib
  Interventions: Drug: camrelizumab + famitinib
- Treatment Arm C (Experimental): famitinib
  Interventions: Drug: famitinib
- Treatment Arm B (Active Comparator): docetaxel
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: camrelizumab + famitinib — camrelizumab for intravenous injection; famitinib malate capsules for oral administration
  Arms: Treatment Arm A
Drug: famitinib — famitinib malate capsules for oral administration
  Arms: Treatment Arm C
Drug: docetaxel — docetaxel for intravenous injection
  Arms: Treatment Arm B

SUMMARY:
This is a randomized, open-label, international, multi-center, phase III trial to evaluate the efficacy, and safety of camrelizumab combined with famitinib malate versus docetaxel as subsequent therapy in Advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic or recurrent non-small cell lung cancer.
2. Failed previous platinum-based chemotherapy and anti-PD-(L)1 monoclonal antibody treatment.
3. Have measurable disease based on RECIST v1.1.
4. ECOG PS score: 0-1.
5. Expected survival ≥ 3 months.
6. Non-surgically sterilized female subjects or women of childbearing potential must be negative for a serum pregnancy test within 3 days prior to the first dose and must be non-lactating. Female subjects of childbearing potential and male subjects with partners of childbearing potential must agree to take highly effective contraceptive measures during the study period and until 6 months after the last study dose.
7. Subjects must participate voluntarily, sign the ICF, have good compliance, and cooperate with follow-up visits.

Exclusion Criteria:

1. Have uncontrolled clinically symptomatic pleural effusion, pericardial effusion, or ascites.
2. Have known history of prior malignancy in the past 3 years.
3. Have active pulmonary tuberculosis.
4. Have clinical symptoms of the heart or heart diseases that are not well controlled.
5. Have hypertension which cannot be well controlled by antihypertensives
6. Urinalysis has indicated that the urine protein is ≥ ++ and quantitative test of urine protein has confirmed that the 24-h urine protein is > 1.0 g.
7. Have a thrombosis tendency or are currently receiving thrombolysis/anticoagulation therapy.
8. Have received major surgery within 4 weeks prior to randomization; or palliative radiotherapy within 2 weeks prior to randomization; or have not recovered from the toxicities and/or complications of previous interventions to NCI-CTCAE Grade ≤ 1.
9. Have known history of arterial/venous thrombosis within 6 months prior to randomization, such as cerebrovascular accidents, deep vein thrombosis and pulmonary embolism.
10. Are currently participating and receiving study therapy or have participated in a study and received the last dose of study drug within 4 weeks (or 5 half-lives of the study drug) prior to randomization.
11. Previous treatment with camrelizumab, docetaxel, and small-molecule VEGFR inhibitors including famitinib.
12. Have other potential factors that may affect the study results or result in the premature discontinuation as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
OS | up to 4 years
  OS is the time interval from the date of randomization to death due to any reason or lost of follow-up.

SECONDARY OUTCOMES:
PFS | up to 4 years
  Progression-Free-Survival, defined as the time from randomization to the first occurrence of disease progression with use of RECIST v1.1 or death from any cause, whichever occurs first.
ORR | up to 4 years
  Objective Response Rate, determined using RECIST v1.1 criteria, defined as best overall response (CR or PR) across all assessment time points.
DoR | up to 4 years
  Duration of Response, determined using RECIST v1.1 criteria.
DCR | up to 4 years
  Disease Control Rate, determined using RECIST v1.1 criteria.
TTF | up to 4 years
  Time to Treatment Failure, defined as the time from randomization to treatment discontinuation.

CONTACTS AND LOCATIONS:
Locations (1):
- Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided